CLINICAL TRIAL: NCT04701164
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of ANX005 in Subjects With Guillain-Barré Syndrome
Brief Title: Efficacy and Safety of ANX005 in Subjects With Guillain-Barré Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANX005-GBS-02
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ANX005 Treatment Group - Dose 1 (Experimental): Participants will receive a single IV infusion of ANX005 (Dose 1) on Day 1.
  Interventions: Drug: ANX005
- ANX005 Treatment Group - Dose 2 (Experimental): Participants will receive a single IV infusion of ANX005 (Dose 2) on Day 1.
  Interventions: Drug: ANX005
- Placebo Group (Placebo Comparator): Participants will receive a single IV infusion of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANX005 — Solution for intravenous infusion
  Arms: ANX005 Treatment Group - Dose 1; ANX005 Treatment Group - Dose 2
Drug: Placebo — Solution for intravenous infusion
  Arms: Placebo Group

SUMMARY:
This study is intended to evaluate the efficacy and safety of ANX005 administered by intravenous (IV) infusion to participants recently diagnosed with Guillain-Barré Syndrome (GBS). The total duration of study participation is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GBS according to the National Institute of Neurological Disorders and Stroke Diagnostic Criteria for Guillain-Barré Syndrome.
* Onset of GBS-related weakness ≤10 days prior to start of infusion.
* GBS-DS score of 3,4, or 5 at screening and at Day 1 prior to infusion.

Exclusion Criteria:

* Clinically significant findings on the screening electrocardiogram (ECG), laboratory test results, or physical examination that are not specific to GBS that may interfere with the conduct of the study, the interpretation of the data, or increase the participant's risk.
* Body weight <30 kilograms (kg) or >150 kg at screening.
* Unresponsive (inexcitable) nerve conduction study results in all nerves tested during screening.
* Previous or intended treatment with either plasma exchange or intravenous immunoglobulin for GBS.
* Diagnosis of a variant of GBS, including Miller Fisher syndrome, Bickerstaff's encephalitis, and overlap syndromes.
* History of prior episode of GBS.
* GBS-related weakness that improved since symptom onset, including an improvement between screening and Day 1 (baseline).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
GBS Disability Score (GBS-DS) at Week 8 | Week 8
Number of Participants with Adverse Events | Through Month 6
  Number participants recently diagnosed with GBS who experience adverse events.

SECONDARY OUTCOMES:
Medical Research Council (MRC) Sum Score at Week 8 | Week 8
MRC Sum Score at Day 8 | Day 8
Duration (Days) of Ventilation Support Over 26 Weeks | 26 weeks
GBS Disability Score (GBS-DS) | Week 26
Number of Participants Requiring Intensive Care Unit Stay | 26 weeks
Duration (Days) of Intensive Care Unit Stays | 26 weeks
Patient Global Impression of Change Scores | Week 8 and Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Annexon, Inc.
Locations (11):
- Bangladesh (2):
  - Dhaka Medical Center, Dhaka
  - National Institute of Neurosciences and Hospital (NINS), Dhaka
- Philippines (9):
  - Baguio General Hospital Medical Center, Baguio City
  - Batangas Medical Center, Batangas
  - Mary Mediatrix Medical Center, Batangas
  - Perpetual Succour Hospital, Cebu City
  - Cotabato Regional Medical Center, Cotabato City
  - Southern Philippines Medical Center, Davao City
  - Jose R. Reyes Memorial Medical Center, Manila
  - West Visayas State University Medical Center, Manila
  - Zamboanga City Medical Center, Zamboanga City

IPD SHARING:
Plan to Share IPD: No